CLINICAL TRIAL: NCT02034058
Title: WEAVE™ Trial: Wingspan StEnt System Post MArket SurVEillance Study
Brief Title: Post Market Surveillance Study of the Wingspan Stent System
Acronym: WEAVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stryker Neurovascular (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: WEAVE Trial
Record Dates: First submitted 2014-01-09; First posted 2014-01-13 (Estimated); Results first posted 2019-12-02 (Actual); Last update posted 2019-12-02 (Actual); Status verified 2019-11

CONDITIONS: Intracranial Atherosclerosis
Keywords: Wingspan Stent System; Wingspan Stent; Intracranial Stent; Ischemic Stroke; Intracranial Atherosclerotic Disease; Intracranial Stenosis
MeSH Terms: conditions — Intracranial Arteriosclerosis; Ischemic Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Wingspan Stent System (Other): Placement of the Wingspan Stent
  Interventions: Device: Wingspan Stent System

INTERVENTIONS:
Device: Wingspan Stent System — The Wingspan Stent System is used with the Gateway PTA Balloon Catheter. The Wingspan Stent System is a self-expanding, Nitinol stent and delivery system intended for use in the treatment of intracranial atherosclerotic disease. The Gateway PTA Balloon Catheter is an over-the-wire balloon catheter intended for the pre-dilation of the lesion prior to insertion and deployment of the Wingspan Stent System.

SUMMARY:
The primary objective of this study is to evaluate the rate of stroke and/or death in patients treated with the Wingspan Stent System, according to the Indications for Use, within 72 hours post procedure.

DETAILED DESCRIPTION:
This research study is a Food and Drug Administration (FDA) mandated post market surveillance study of the Wingspan® Stent System, also known as the WEAVE™ Trial. The purpose of this trial is to fulfill a FDA requirement to evaluate the rate of stroke and/or death within 72 hours of the procedure, in patients who have a Wingspan Stent implanted in accordance with the Indications for Use.

ELIGIBILITY:
All patients for whom treatment with the Wingspan Stent System is considered.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2013-12; Primary Completion 2019-08 (Actual); Study Completion 2019-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Alexander, M.D., Principal Investigator — Cedars-Sinai Medical Center; Wengui Yu, M.D., Principal Investigator — University of California, Irvine
Locations (26):
- United States (26):
  - University of Alabama-Birmingham, Birmingham, Alabama
  - Sutter Eden Medical Center, Castro Valley, California
  - Southern California Permanente Medical Group, Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - UCSD Medical Center, San Diego, California
  - Santa Barbara Cottage Hospital, Santa Barbara, California
  - Mount Sinai Medical Center, Miami Beach, Florida
  - Emory University, Grady Memorial Hospital, Atlanta, Georgia
  - WellStar Health System, Marietta, Georgia
  - University of Chicago, Chicago, Illinois
  - Cadence Health, Northwestern Medicine Central DuPage Hospital, Winfield, Illinois
  - Baptist Health Lexington, Lexington, Kentucky
  - University of Kentucky Medical Center, Lexington, Kentucky
  - University of Massachusetts, Worcester, Worcester, Massachusetts
  - St. John Hospital and Medical Center, Inc., Detroit, Michigan
  - SSM DePaul Health Center, Bridgeton, Missouri
  - Columbia University Medical Center, New York, New York
  - University Hospital of Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Tennessee Interventional Associates, Chattanooga, Tennessee
  - Valley Baptist Harlingen, Harlingen, Texas
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - University of Washington, Harborview Medical Center, Seattle, Washington
  - Multicare Medical Center, Tacoma, Washington

REFERENCES:
- [Derived] Alexander MJ, Zauner A, Chaloupka JC, Baxter B, Callison RC, Gupta R, Song SS, Yu W; WEAVE Trial Sites and Interventionalists. WEAVE Trial: Final Results in 152 On-Label Patients. Stroke. 2019 Apr;50(4):889-894. doi: 10.1161/STROKEAHA.118.023996. PMID 31125298

RESULTS

PARTICIPANT FLOW:
Groups:
- Stenting: Prospective, single-arm, consecutive enrollment, post market surveillance study of patients treated with the Wingspan Stent System, according to the Indications for Use.
Period: Overall Study
Arm/Group | Stenting
Started | 152 (Study stopped early per pre-defined criteria for interim analysis.)
Completed | 149
Not Completed | 3
Not completed — Death | 3

BASELINE CHARACTERISTICS:
Groups:
- Stenting: Prospective, single-arm, consecutive enrollment, post market surveillance study of patients who have a Wingspan stent procedure attempted.
Arm/Group | Stenting
Number analyzed (Participants) | 152
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.89 (10.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 71
  Male | 81
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: Caucasian | 101
  Race/Ethnicity: African American or Black | 30
  Race/Ethnicity: Asian | 4
  Race/Ethnicity: Hispanic or Latino | 12
  Race/Ethnicity: Multiracial | 5
Baseline modified Rankin Scale [Count of Participants; unit: Participants] — mRS scale is as follows: 0 - No symptoms. 1 - No significant disability. Able to carry out all usual activities, despite some symptoms. 2 - Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities. 3 - Moderate disability. Requires some help, but able to walk unassisted. 4 - Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted. 5 - Severe disability. Requires constant nursing care and attention, bedridden, incontinent" or similar).
  Participants
    0 | 20
    1 | 37
    2 | 52
    3 | 43
    4 | 0
    5 | 0

OUTCOME MEASURES:

1. Primary Outcome: Rate of Stroke or Death Among Participants
Description: The primary endpoint in this study is the rate of stroke (ischemic or hemorrhagic) or death within 72 hours of the procedure. Ischemic stroke was defined as a neurological deficit that is thought to have an ischemic cause and is detectable on examination at least 24 hours after onset of symptoms. Hemorrhagic stroke was defined as a symptomatic intracerebral, subarachnoid, or primary intraventricular hemorrhage. The type of stroke was confirmed by imaging.
Time Frame: within 72 hours of the procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Stenting
Number analyzed (Participants) | 152
Participants | 4

2. Secondary Outcome: Rate of Ischemic Stroke Among Participants
Description: Ischemic stroke was defined as a neurological deficit that is thought to have an ischemic etiology and is detectable on examination at least 24 hours after onset of symptoms.
Time Frame: within 72 hours post procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Stenting
Number analyzed (Participants) | 152
Participants | 1

3. Secondary Outcome: Rate of Neurological Death Among Participants
Description: A diagnosis of death by neurological criteria
Time Frame: within 72 hours post procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Stenting
Number analyzed (Participants) | 152
Participants | 2

4. Secondary Outcome: Rate of Stroke Recovery Among Participants
Description: Stroke recovery at 90 days post procedure is defined by return to baseline mRS at Day 90.
Time Frame: at 90 days post procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Stenting
Number analyzed (Participants) | 152
Participants | 0

5. Secondary Outcome: Rate of Stroke in the Territory of the Stented Artery Among Participants
Description: Stroke in the vascular territory of the stented artery
Time Frame: within 72 hours post procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Stenting
Number analyzed (Participants) | 152
Participants | 4

ADVERSE EVENTS:
Time Frame: Serious and Other Adverse Events were monitored/assessed for up to 72 hours post-procedure. All-Cause Mortality was monitored/assessed through 90 days post procedure.
Description: Only neurological AEs, bleeding/hemorrhagic AEs (including non-neurological events), groin puncture AEs and AEs that resulted in death experienced by the study subject after enrollment were collected.
Arm/Group | Stenting
All-Cause Mortality (participants affected / at risk) | 3/152
Serious Adverse Events (participants affected / at risk) | 9/152
Other Adverse Events (participants affected / at risk) | 12/152
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stenting (N=152)
Haemorrhagic stroke (Nervous system disorders) | 3 (3)
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 1 (1)
Neurological decompensation (Nervous system disorders) | 1 (1)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stenting (N=152)
Administration site pain (General disorders) | 2 (2)
Application site haematoma (General disorders) | 3 (3)
Haemorrhage intracranial (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 3 (3)
Muscular weakness (Nervous system disorders) | 1 (1)
Neurological symptom (Nervous system disorders) | 2 (2)
Transient ischaemic attack (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-10-13): https://cdn.clinicaltrials.gov/large-docs/58/NCT02034058/Prot_SAP_000.pdf